CLINICAL TRIAL: NCT06728969
Title: A Prospective Comparative Study to Evaluate a Novel Algorithm Using Data Derived from a Non-Invasive Digital Biomarker As a Diagnostic Aid for ADHD in Youth Ages 6-17.
Brief Title: A Comparative Study to Evaluate a Novel Algorithm As a Diagnostic Aid for ADHD in Youth Ages 6-17.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MindTension (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-0000
Record Dates: First submitted 2024-11-23; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-11

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: The study will include a group of subjects who have ADHD and subjects who are healthy controls based on the specialist clinician assessment.
  Following the specialist clinician assessment each subject will undergo a test using the FDA cleared T.O.V.A and MindTension's MT1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- ADHD group (Experimental): Subjects will be evaluated for ADHD using clinically established reference standard interviews and psychometric tools with demonstrated validity, including the K-SADS and ADHD-RS-5, in accordance with DSM-5 criteria. IQ will be estimated using two subtests of the WASI.
  Interventions: Device: MT1 Auditory startle response patterns analysis algorithm; Device: T.O.V.A. Continuous Performance Test
- Non-ADHD group (Experimental): Subjects will be evaluated using clinically established reference standard interviews and psychometric tools with demonstrated validity, including the K-SADS and ADHD-RS-5, in accordance with DSM-5 criteria. IQ will be estimated using two subtests of the WASI.
  Interventions: Device: MT1 Auditory startle response patterns analysis algorithm; Device: T.O.V.A. Continuous Performance Test

INTERVENTIONS:
Device: MT1 Auditory startle response patterns analysis algorithm — Objective measurements of attention and inhibition.
Device: T.O.V.A. Continuous Performance Test — Objective measurements of attention and inhibitory control.

SUMMARY:
This study aims to demonstrate the accuracy of the MT1 algorithm using the MindTension biometric sensor device as a diagnostic aid for healthcare providers in diagnosing ADHD in youth ages ≥ 6 to ≤17 years.

DETAILED DESCRIPTION:
The study aims to demonstrate the accuracy of the MT1 algorithm. The output of the MT1 algorithm will be compared to a Gold Standard clinical diagnosis made by specialist clinician diagnosis supported by the Kiddie SADS Present and Lifetime semi-structured interview (K-SADS-PL) and norm-referenced measures of current ADHD symptom frequency and severity using the ADHD-RS-5 rating scale. Diagnosis will be scaled according to the Diagnostic and Statistical Manual of Mental Disorders- 5 (DSM-5) criteria, and made with agreement between two licensed specialists in ADHD (a Clinical Psychologist and a Psychiatrist).

Further to the above, demonstrate that the agreement between the MT1 output and the specialist clinician diagnosis will be non-inferior to the level of agreement between the clinician diagnosis with the Test of Visual Attention (TOVA) FDA cleared device.

ELIGIBILITY:
Inclusion Criteria:

1. Parent provision of signed and dated informed consent form
2. Child stated willingness to comply with all study procedures and availability for the duration of the study
3. Any gender, aged 6 to 17 years
4. Stimulant naïve or willing to wash out of stimulant for 3 days (approximately 72 hours) prior to testing with biometric and performance devices (MindTension + TOVA)
5. ADHD Group: Diagnosed with symptoms consistent with ADHD as determined by Mini Kid + an ADHD-RS score of 1.5SD above mean for age and sex
6. Control group: No diagnosable disorder on the Mini kid, and an ADHD-RS score within 1SD of the mean for age and sex.

Exclusion Criteria:

1. Current use of psychotropic medications that cannot be washed out in 3 days (approximately 72 hours)
2. Known current seizure disorder (history of febrile seizure allowed).
3. Presence of specific devices (e.g., cardiac pacemaker) that may interfere with the MindTension monitor
4. IQ<70 by clinician judgment
5. Meeting FULL criteria for current PTSD, GAD, MDD, or any lifetime diagnosis of ASD, Bipolar disorder, or psychotic disorder that was, in the opinion of the investigator, correctly obtained. May have symptoms of anxiety or dysthymia/depression not meeting criteria for a full disorder, or disorders such as simple phobia
6. Deaf or hearing impaired, since this will make it difficult to hear and respond to the auditory stimuli.
7. Inability to complete the assessments.
8. Any other concerns in the judgment of the PI.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2024-06-02 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Overall Agreement Rate (OAR) - probability that the test will be normal and the condition is normal or positive and the condition is positive, out of all subjects. | From the beginning of clinical assessment until the end of testing (approximately 1-2 days).
  The outcome measure will be calculated by using the following formula:
  Over All Agreement = (True Positive + True Negative) / (True Positive + True Negative + False Positive + False Negative) X 100.

SECONDARY OUTCOMES:
Positive Predicted Value (PPV) - conditional probability that the condition will be positive if the test is positive. | From the beginning of clinical assessment until the end of testing (approximately 1-2 days).
  The outcome measure will be calculated using the following formula:
  Positive Predicted Value = (True Positive) / (True Positive + False Positive) X 100
Negative Predicted Value (NPV) - conditional probability that the condition will be normal if the test is normal. | From the beginning of clinical assessment until the end of testing (approximately 1-2 days).
  The outcome measure will be calculated using the following formula:
  Negative Predicted Value = (True Negative) / (True Negative + False Negative) X 100
Sensitivity - conditional probability that the test will be positive if the condition is positive. | From the beginning of clinical assessment until the end of testing (approximately 1-2 days).
  The outcome measure will be calculated using the following formula:
  Sensitivity = (True Positive) / (True Positive + False Negative) X 100
Specificity - conditional probability that the test will be normal if the condition is normal. | From the beginning of clinical assessment until the end of testing (approximately 1-2 days).
  The outcome measure will be calculated using the following formula:
  Specificity = (True Negative) / (True Negative + False Positive) X 100

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Newcorn, MD Professor, Principal Investigator — Director, Division of ADHD and Learning Disorders Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States